## **Evaluation of the Clinical and Radiographic Success of Platelet-Rich Fibrin, Chitosan,** and Blood Clot as Scaffolds in Regenerative Endodontic Treatment of Molars

NCT ID not yet assigned

**Document Date: 10.01.2022** 

## INFORMED VOLUNTARY CONSENT FORM

We invite you to the study titled "Evaluation of Clinical and Radiological Success of the Platelet-Rich Fibrin, Chitosan and Blood Clot as a Scaffold in the Regenerative Endodontic Treatment of Molar Teeth" conducted by ....... Before you decide whether to take part in this study, you need to know why and how it will be conducted. Therefore, it is very important that you read and understand this form. You can choose whether or not to take part in this study. If you don't understand something or if you need more information, please ask us. You have the right to choose not to be in the study or to leave the study at any time after you join. You won't be punished if you leave the study, and you can choose to stop participating or withdraw from the study without losing any rights. If new information comes up about the research that could affect the volunteer's decision to keep participating, the volunteer or their legal representative will be told right away. The information you provide on these forms will only be used for the research. Even if the research is published, your name and other personal information will remain strictly confidential and will not be shared with anyone else. If we collect your biological materials (like blood, urine, tissue, etc.), we will give you information about what the materials are, why we collected them, and where we will analyze them (if we analyze them abroad, we will tell you where the materials will be sent). The Informed Consent Form we have prepared does not contain any information that would eliminate the legal rights of the volunteer or legal representative. It also does not contain any information that would relieve the researcher, institution, sponsor, or their representatives from any liability arising from their own negligence.

The legal guardians or guardians of the participants/volunteers under the age of 18 were given the necessary explanations and were informed. The study was approved. If you take part in the study and answer the questions, you are giving your permission to take part in the research. Don't feel pressured or influenced by anyone when answering the questions on the forms.

- 1. Full name of the study: The study "Evaluation of Clinical and Radiological Success of the Platelet-Rich Fibrin, Chitosan and Blood Clot as a Scaffold in the Regenerative Endodontic Treatment of Molar Teeth"
- 2. Did you tell the volunteer that the study was a study? Yes.
- 3. What is the purpose of the study? The study compares the effects of three different materials used as "scaffolds" in regenerative endodontic treatment. The materials are compared in terms of their clinical and radiographic effects.
- 4. How long do you think the volunteer will need to continue the study? It will take between 12 and 18 months.
- 5. How many volunteers do you think will participate in the study? There are at least 24 teeth.
- 6. If there are any, what treatments will be used in the study? Regenerative Endodontic Treatment

- 7. If so, is there a way to randomly assign volunteers to research groups for different treatments? There is no difference in treatment. The clinic will keep records of the treatment given and do a statistical evaluation. You will not be given any more appointments or X-rays as part of this study.
- 8. Explain all methods to be followed or applied to the volunteer, including invasive methods to be applied during the research, in terms that the volunteer can understand. After the dentist numbs the tooth, they will clean and fill the tooth with medicine and close it with a temporary filling. In the second session, the temporary filling will be removed, and the canals will be washed again. Then, various materials will be placed in the canals to help the roots grow. After the dentist puts in the materials, the tooth will be filled. A special metal coating (stainless steel crown) will be applied to teeth that are too damaged to be filled. Then, we will check the tooth every three months to see how it is healing.
- 9. Explain the experimental parts of the research: The experimental part of this study is to compare the long-term success of materials that have been shown to be successful in previous studies on molar teeth.
- 10. Explain the expected risks or discomforts that the volunteer may face (including the expected risks or discomforts that the embryo, fetus, or infants may face if the research is conducted on pregnant or postpartum women): None.
- 11. If there is no clinical benefit for the volunteer, will they be informed about this situation? Yes.
- 12. Explain the other ways to treat the volunteer and the possible good and bad points of each method. Apexification treatments can also be used on teeth with unclosed root tips. However, these treatments only close the root tip without increasing its thickness or length. So, it's not the preferred method anymore. Another treatment option for immature necrotic teeth is root canal treatment after apical occlusion with MTA. Another benefit of this method is that it's a one-time deal. The root thickness and length don't increase; only the root tip is closed. So, it's not recommended unless it's absolutely necessary. It is preferred in patients who cannot continue treatment because of the number of sessions. Regeneration, which was used in the study, is also the most recommended and applied method in the literature today.
- 13. If necessary, the volunteer will be given the compensation and/or treatment they are owed. The necessary expenses will be covered according to the relevant legislation.
- 14. What are the volunteers' responsibilities? Have you written a list of the things you need and had the volunteer sign it? Volunteers must regularly visit check-up locations and follow oral hygiene rules. Information was given on these issues, and signatures were obtained.

## CONSENT TO PARTICIPATE IN THE RESEARCH

I have read all the explanations in the informed consent form and explained them to my child in a way that he/she can understand. The doctor explained the research to me in writing and verbally. The purpose and subject of the research are stated above. I know that my child can stop participating in the research at any time, and they don't have to give a reason. I, as a mother or father or legal guardian, agree to my child's choice to take part in the research. I agree to this without feeling pressured or forced.

PARENT/GUARDIAN (If applicable)

NAME-SURNAME

**SIGN** 

| ADRESS | _ |
|-------------------------|------|
| PHONE NUMBER | |
| DATE | - |
| RESEARCHER | SIGN |
| NAME-SURNAME and DEGREE | |
| ADRESS | |
| PHONE NUMBER | |
| DATE | |